CLINICAL TRIAL: NCT04288934
Title: Assessment of Safety and Effectiveness of Mesenchymal Stem Cells in the Treatment of Spinal Cord Injury (SCI) Patients.
Brief Title: Treatment of Spinal Cord Injuries With (AutoBM-MSCs)vs (WJ-MSCs).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Head of Neuroscience Research, University of Jordan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCICTC
Record Dates: First submitted 2019-09-23; First posted 2020-02-28 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injuries; Mesenchymal Stem Cells; Allogenic; Bone marrow derived Mesenchymal stem cells; American Spinal Injury Association Impairment Scale
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Patients with complete transection of the spinal cord. Each group will then be subdivided into 2 subgroups with of 5 patients each; the 1st subgroup will be the patients with chronic SCI and the 2nd subgroup will be for the patients with subacute SCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with complete transection of the spinal cord (Active Comparator): This group of patients with complete transection of the spinal cord group will then be subdivided into 2 subgroups with of 5 patients each; the 1st subgroup will be the patients with chronic SCI and the 2nd subgroup will be for the patients with subacute SCI. All patients will receive AutoBM-MSCs by a specialized spine surgeon into the spinal medulla.
  Interventions: Biological: Collection and expansion of BM-MSC; Diagnostic Test: VI-SCI evaluation and patients' follow up
- patients with SCI without total transaction. (Active Comparator): This group will then be subdivided into 2 subgroups with of 5 patients each; the 1st subgroup will be the patients with chronic SCI and the 2nd subgroup will be for the patients with subacute SCI. All patients will receive WJ-MSCs by a specialized spine surgeon into the spinal medulla.
  Interventions: Biological: Collection and expansion of BM-MSC; Diagnostic Test: VI-SCI evaluation and patients' follow up

INTERVENTIONS:
Biological: Collection and expansion of BM-MSC — MSCs collection from patients owns marrow using a volume of 20 ml of bone marrow obtained from iliac crest of SCI patients under local anesthesia. Manipulations of blood and bone marrow are to be done according to Good Laboratory Practice (GLP) using the gradient sedimentation method.
Diagnostic Test: VI-SCI evaluation and patients' follow up — * At 6, and 12 months post MSCs transplantation, patients' spine will be imaged using 3 Tesla MRI and compared to baseline.
  * The (ASIA)/(ISNCSCI) score will be repeated every 3 months to evaluate any motor or neurological changes
  * The Spinal Cord Independence Measure (SCIM III) score will be repeated every 3 months to evaluate the effect on daily activities.
  * Blood samples will be withdrawn from patients at 3 months interval for biomarkers detection.

SUMMARY:
This study aims to assess and compare the safety and effectiveness of Autologous Bone Marrow-Derived MSCs (AutoBM-MSCs) in one group(group A) of SCI who are unlikely to be able to walk independently without treatment after 1 year of SCI, in the other group (group B) to assess the second group of Wharton Jelly derived mesenchymal stem cells ( WJ-MSCs) in the treatment of acute and subacute spinal cord injury (SCI) patients.

DETAILED DESCRIPTION:
The study will be directed by the Cell Therapy Center (CTC) in Jordan, where 20 SCI patients meeting the inclusion criteria will be recruited and divided according to the type of injury into two groups; Group A for patients with complete transection of the spinal cord, and Group B for SCI without a total transaction,10 patients will receive (AutoBM-MSCs)and the other 10 patients with acute and subacute spinal cord injury will receive(WJ-MSCs) by a specialized spine surgeon into the spinal medulla. The outcomes and improvements will be assessed using the American Spinal Injury Association (ASIA) Impairment Scale (AIS) and the Spinal Cord Independence Measure (SCIM) version III, in addition to blood tests, MRI, and somatosensory evoked potential (SSEP).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Complete SCI grade AIS-A or -B, or incomplete C
* SCI between cervical levels C5 and thoracic level T11
* At least 12 weeks since time of injury
* Prediction rule score of 10 or less
* Cognitively unaffected
* Motivated for stem cell transplantation

Exclusion Criteria:

* Reduced cognition
* Age under 18 years or above 70 years
* Significant osteoporosis in spine and/or joints
* Pregnancy (Adequate contraceptive use is required for women in fertile age)
* Anoxic brain injury
* Neurodegenerative diseases
* Evidence of meningitis
* Positive serology for HIV, HBV, HCV, or Syphilis.
* Medical Complications that contraindicate surgery, including major respiratory complications.
* Use of metal implants close to vascular structures (such as cardiac pacemaker or prosthesis) that contraindicate MRI.
* Other medical conditions which can interfere with stem cell transplantation
* Inability to provide informed consent.
* Uncorrected vision
* Cardiac abnormalities and uncontrolled hypertension

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
SCI evaluation and patients follow up | 3 months
  the (ASIA)/(ISNCSCI) to evaluate any motor or neurological changes, and the spinal cord independence measure (SCIM III) score to evaluate the effect on daily activities .these tests will be repeated every 3 months.
  blood samples will be withdrawn from patients as well to detect any biomarkers.
SCI evaluation and MSCs transplantation | 6-12 months
  post MSCs transplantation, patients' spine will be imaged using 3 Tesla MRI and compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Center, University of Jordan, Amman, Jordan